CLINICAL TRIAL: NCT03044574
Title: Trial to Assess the Effectiveness of Intermittent Pneumatic Compression in the Prevention of Postoperative Venous Thromboembolism in Surgical Patients at Extremely High Risk
Brief Title: Intermittent Pneumatic Compression in Surgical Patients at Extremely-high Risk for Venous Thromboembolism
Acronym: IPCSUPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pirogov Russian National Research Medical University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Kirill Lobastov, Associated Professor, Pirogov Russian National Research Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IPCSUPER
Record Dates: First submitted 2017-02-01; First posted 2017-02-07 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2020-04

CONDITIONS: Venous Thromboembolism; Venous Thrombosis
Keywords: venous thromboembolism; deep vein thrombosis; pulmonary embolism; prevention; intermittent pneumatic compression; sequential pneumatic compression; surgery; elastic compression; low-molecular weight heparin; prophylaxis
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Intervention Model Description: A randomized clinical study to assess efficacy and safety of intermittent pneumatic compression device (SCD) application in combined prevention of postoperative VTE in surgical patients at high and extremely high risk receiving graduated compression stockings and early/delayed prophylactic anticoagulation with low-molecular weight heparins.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Experimental group (SCD + GCS + LMWH) (Experimental): SCD: Intermittent pneumatic compression (IPC) with Kendall SCD™ Sequential Compression System 700 used continuously when the patient is in bed with 6-hours night interval free of compression: from 0 a.m. to 6 a.m. In the ICU SCD used continuously all day, and in surgery department - all time of bed resting. SCD used until discharge.
  GCS: Thigh-length graduated compression stockings with pressure of 18-21 mm. Hg at the ankle used all the time until discharge plus one month after discharge
  LMWH: LMWH enoxaparin (Clexane) 40 mg once a day subcutaneously started on 1st or 2-5th postoperative day according to the bleeding risk and used until discharge.
  Interventions: Device: SCD; Device: GCS; Drug: LMWH
- Control group (GCS + LMWH) (Active Comparator): GCS: Thigh-length graduated compression stockings with pressure of 18-21 mm. Hg at the ankle used all the time until discharge plus one month after discharge
  LMWH: LMWH enoxaparin (Clexane) 40 mg once a day subcutaneously started on 1st or 2-5th postoperative day according to the bleeding risk and used until discharge.
  Interventions: Device: GCS; Drug: LMWH

INTERVENTIONS:
Device: SCD — Intermittent pneumatic compression (IPC) with Kendall SCD™ Sequential Compression System 700 used continuously when the patient is in bed with 6-hours night interval free of compression: from 0 a.m. to 6 a.m. In the ICU SCD used continuously all day, and in surgery department - all time of bed resting. SCD used until discharge.
  Arms: Experimental group (SCD + GCS + LMWH)
Device: GCS — Thigh-length graduated compression stockings with pressure of 18-21 mm. Hg at the ankle used all the time until discharge plus one month after discharge
Drug: LMWH — LMWH enoxaparin (Clexane) 40 mg once a day subcutaneously started on 1st or 2-5th postoperative day according to the bleeding risk and used until discharge.

SUMMARY:
The aim of the study is to evaluate efficacy and safety of venous thromboembolism prophylaxis by the combination of graduated compression stockings (GCS), standard doses of low-molecular-weight heparins (LMWH) and sequential compression device (SCD) in the mixed group of surgical patients at high and extremely high risk for venous thromboembolism.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is the most common complication after major surgery, especially in high-risk patients. But the high-risk group is inhomogeneous. Some patients included in this group have an extremely high prevalence of postoperative venous thrombosis and pulmonary embolism, in whom the standard complex prophylaxis with elastic compression and standard anticoagulation is less effective. This is particularly so, in patients having a Caprini score of 11 and more, so that at the background of standard prophylaxis postoperative DVT is 10 times higher. This group of patients needs a more effective protocol for VTE prevention.

Sequential compression devices (SCD) combined with graduated elastic compression stockings (GCS) or without them were found to be effective in the prevention of VTE in high-risk patients, especially after neurosurgical interventions, even without the administration of anticoagulants. However, their efficacy in patients at "extremely high risk", having 11+ Caprini scores has not been assessed yet. The aim of the current study is to evaluate efficacy and safety of VTE prophylaxis by the combination of graduated compression stockings (GCS), standard doses of low-molecular-weight heparins (LMWH) and sequential compression device (SCD) in the mixed group of surgical patients at high and extremely high risk for venous thromboembolism

The expected outcome of the study is a reduction of asymptomatic postoperative venous thrombosis rate in the hospital and reduction in all VTE during 6 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age over 40
* Major surgery undergone*
* High risk of postoperative VTE according to a National guideline**
* 11+ Caprini scores
* Informed consent is given

Exclusion Criteria:

* Acute deep vein thrombosis (DVT) at baseline
* Performed inferior vena cava (IVC) plication or implanted IVC filter
* Regular preoperative anticoagulation
* Postoperative anticoagulation needed at therapeutic doses
* Absence of anticoagulation for more than 5 days after surgery
* Coagulopathy (not related to Disseminated intravascular coagulation syndrome)
* Thrombocytopenia
* Hemorrhagic diathesis
* Lower limb soft tissue infection
* Ankle-brachial index < 0.6

  * Major surgery - intervention under endotracheal anesthesia with duration of more than 60 min.

    * In accordance with a standard stratification system, high risk of VTE group includes patients over 60 years old after major surgery and patients 40-60 years old with additional risk factors after major surgery.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirill Lobastov, PhD, Principal Investigator — Pirogov Russian National Research Medical University
Locations (2):
- Russia (2):
  - Clinical Hospital no.1 of the President's Administration of Russian Federation, Moscow
  - Moscow Clinical Hospital no.24, Moscow

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schastlivtsev I, Lobastov K, Barinov V, Kanzafarova I. Diosmin 600 in adjunction to rivaroxaban reduces the risk of post-thrombotic syndrome after femoropopliteal deep vein thrombosis: results of the RIDILOTT DVT study. Int Angiol. 2020 Oct;39(5):361-371. doi: 10.23736/S0392-9590.20.04356-4. Epub 2020 Apr 29. PMID 32348101
- [Derived] Lobastov K, Sautina E, Alencheva E, Bargandzhiya A, Schastlivtsev I, Barinov V, Laberko L, Rodoman G, Boyarintsev V. Intermittent Pneumatic Compression in Addition to Standard Prophylaxis of Postoperative Venous Thromboembolism in Extremely High-risk Patients (IPC SUPER): A Randomized Controlled Trial. Ann Surg. 2021 Jul 1;274(1):63-69. doi: 10.1097/SLA.0000000000004556. PMID 33201130

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The total amount of 812 patients were screened during the enrollment period, 405 of them were excluded: Caprini score of <11 (n=304); a various regimen of anticoagulation (n=48); venous thrombosis at the baseline (n=31); declined participation (n=18); implanted inferior vena cava filter (n=4).
Groups:
- Experimental Group (SCD + GCS + LMWH): Sequential Compression Device (SCD): Intermittent pneumatic compression (IPC) with Kendall SCD™ Sequential Compression System 700 used continuously when the patient is in bed with 6-hours night interval free of compression: from 0 a.m. to 6 a.m. In the ICU SCD used continuously all day, and in surgery department - all time of bed resting. SCD used until discharge.
  Graduated Compression Stockings (GCS): Thigh-length graduated compression stockings with pressure of 18-21 mm. Hg at the ankle used all the time until discharge plus one month after discharge
  Low-Molecular-Weight-Heparin (LMWH): LMWH enoxaparin (Clexane) 40 mg once a day subcutaneously started on 1st or 2-5th postoperative day according to the bleeding risk and used until discharge.
Period: Overall Study
Arm/Group | Experimental Group (SCD + GCS + LMWH) | Control Group (GCS + LMWH)
Started | 204 | 203
Inpatient Period | 204 | 203
30 Days After Surgery | 193 | 194
180 Days After Surgery | 167 | 158
Completed | 167 | 158
Not Completed | 37 | 45
Not completed — Lost to Follow-up | 37 | 45

BASELINE CHARACTERISTICS:
Groups:
- Experimental Group (SCD + GCS + LMWH): Sequential Compression Device (SCD): Intermittent pneumatic compression (IPC) with Kendall SCD™ Sequential Compression System 700 used continuously when the patient is in bed with a 6-hours night interval free of compression: from 0 a.m. to 6 a.m. In the ICU SCD used continuously all day, and in the surgery department - all time of bed rest. SCD used until discharge.
  Graduated Compression Stockings (GCS): Thigh-length graduated compression stockings with a pressure of 18-21 mm. Hg at the ankle used all the time until discharge plus one month after discharge
  Low-Molecular-Weight Heparin: LMWH enoxaparin (Clexane) 40 mg once a day subcutaneously started on 1st or 2-5th postoperative day according to the bleeding risk and used until discharge.
- Total: Total of all reporting groups
Arm/Group | Experimental Group (SCD + GCS + LMWH) | Control Group (GCS + LMWH) | Total
Number analyzed (Participants) | 204 | 203 | 407
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (9.6) | 68.8 (10.0) | 68.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 118 | 247
  Male | 75 | 85 | 160
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 204 | 203 | 407
Surgical profile [Count of Participants; unit: Participants] — Abdominal surgery suggests oned and laparoscopic interventions of abdominal cavity and abdominal wall. Non-abdominal surgery contains open and endoscopic interventions on thoracic cavity and thoracic wall, head, and neck, gynecological and urological pelvic surgery, intracranial surgery
  Participants
    Addominal surgery | 131 | 147 | 278
    Non-abdominal surgery | 73 | 56 | 129
Malignancy [Count of Participants; unit: Participants] — Malignancy suggests that patients required surgery due to verified (previously or intraoperatively) malignant tumor
  Participants | 171 | 165 | 336
Caprini score [Mean (Standard Deviation); unit: units on a scale] — Caprini score is a combination of 39 individual risk factors for postoperative venous thromboembolism (VTE), evaluated from 1 to 5 scores. The total amount of scores ranges from 0 to 87: score of 0 suggests the very low risk for VTE; a score of 1-2 suggests the low risk for VTE; a score of 3-4 suggests the intermediate risk for VTE; a score of 5-10 suggests the high fisk for VTE and a score of 11 and higher suggests the extremely high risk for VTE. Patients will a score of 11 and higher represent the target population for the current trial.
  units on a scale | 11.5 (1.8) | 11.4 (1.9) | 11.4 (1.9)
Number of patients with Caprini score of 11 and higher [Count of Participants; unit: Participants] — Caprini score is a combination of 39 individual risk factors for postoperative VTE, evaluated from 1 to 5 scores. The total amount of scores ranges from 0 to 87: score of 0 suggests the very low risk for VTE; a score of 1-2 suggests the low risk for VTE; a score of 3-4 suggests the intermediate risk for VTE; a score of 5-10 suggests the high fisk for VTE and a score of 11 and higher suggests the extremely high risk for VTE. Patients will a score of 11 and higher represent the target population for the current trial.
  Participants | 145 | 140 | 285

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Asymptomatic Venous Thrombosis of Lower Limbs as Detected by Duplex Ultrasound
Description: Asymptomatic deep and/or superficial vein thrombosis of lower limbs detected by duplex ultrasound performed at baseline and then every 3-5 days after surgery until discharge.
Time Frame: time of discharge from the hospital or death, up to 45 days
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group (SCD + GCS + LMWH) | Control Group (GCS + LMWH)
Number analyzed (Participants) | 204 | 203
Participants | 1 | 34
Statistical Analysis 1: Comparison: Experimental Group (SCD + GCS + LMWH) vs Control Group (GCS + LMWH); Test type: Superiority; p < 0.001, Fisher Exact

2. Secondary Outcome: Number of Patients With Proximal Deep Venous Thrombosis as Detected by Duplex Ultrasound
Description: Proximal deep vein thrombosis defined as thrombus of popliteal, femoral, iliac veins and/or inferior vena cava. Detected by duplex ultrasound performed at baseline and then every 3-5 days after surgery until discharge.
Time Frame: time of discharge from the hospital or death, up to 45 days
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group (SCD + GCS + LMWH) | Control Group (GCS + LMWH)
Number analyzed (Participants) | 204 | 203
Participants | 0 | 5
Statistical Analysis 1: Comparison: Experimental Group (SCD + GCS + LMWH) vs Control Group (GCS + LMWH); Test type: Superiority; p = 0.03, Fisher Exact

3. Secondary Outcome: Number of Patients With Isolated Calf Muscle Vein Thrombosis as Detected by Duplex Ultrasound
Description: Isolated calf muscle vein thrombosis was defined as thrombosis of soleal, gastrocnemius or other calf muscle veins not extended into tibial, or peroneal, or popliteal veins. Detected by duplex ultrasound performed at baseline and then every 3-5 days after surgery until discharge.
Time Frame: time of discharge from the hospital or death, up to 45 days
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group (SCD + GCS + LMWH) | Control Group (GCS + LMWH)
Number analyzed (Participants) | 204 | 203
Participants | 1 | 15
Statistical Analysis 1: Comparison: Experimental Group (SCD + GCS + LMWH) vs Control Group (GCS + LMWH); Test type: Superiority; p < 0.001, Fisher Exact

4. Secondary Outcome: Number of Patients With Pulmonary Embolism
Description: Symptomatic pulmonary embolism (PE) that occurred during the inpatient period of treatment and confirmed by computed tomography pulmonary angiogram (CTPA) or single-photon emission computed tomography with computed tomography (SPECT/CT) or autopsy
Time Frame: time of discharge from the hospital or death, up to 45 days
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group (SCD + GCS + LMWH) | Control Group (GCS + LMWH)
Number analyzed (Participants) | 204 | 203
Participants | 0 | 5
Statistical Analysis 1: Comparison: Experimental Group (SCD + GCS + LMWH) vs Control Group (GCS + LMWH); Test type: Superiority; p = 0.03, Fisher Exact

5. Secondary Outcome: Number of Patients Died From Any Reason
Description: Inpatient postoperative mortality: number of patients died from any reason during the inpatient period of treatment
Time Frame: time of discharge from the hospital or death, up to 45 days
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group (SCD + GCS + LMWH) | Control Group (GCS + LMWH)
Number analyzed (Participants) | 204 | 203
Participants | 6 | 10
Statistical Analysis 1: Comparison: Experimental Group (SCD + GCS + LMWH) vs Control Group (GCS + LMWH); Test type: Superiority; p > 0.05, Fisher Exact

6. Secondary Outcome: Number of Patients With Leg Skin Injury
Description: Leg skin injury defined as any skin hyperemia, maceration, laceration, bubbles, erosion or ulceration in the zone of application for GCS and SCD on the lower limbs revealed by clinical inspection of the skin and soft tissues until discharge
Time Frame: time of discharge from the hospital or death, up to 45 days
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group (SCD + GCS + LMWH) | Control Group (GCS + LMWH)
Number analyzed (Participants) | 204 | 203
Participants | 25 | 15
Statistical Analysis 1: Comparison: Experimental Group (SCD + GCS + LMWH) vs Control Group (GCS + LMWH); Test type: Superiority; p > 0.05, Fisher Exact

7. Secondary Outcome: Number of Patients With Symptomatic and Asymptomatic VTE Events at 30 Days After Surgery
Description: Taking into account all VTE events: asymptomatic revealed by duplex ultrasound, symptomatic confirmed by duplex ultrasound, CTPA, SPECT/CT, autopsy in patients discharged from the hospital and still receiving inpatients care at 30 days after surgery.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group (SCD + GCS + LMWH) | Control Group (GCS + LMWH)
Number analyzed (Participants) | 193 | 194
Participants | 1 | 35
Statistical Analysis 1: Comparison: Experimental Group (SCD + GCS + LMWH) vs Control Group (GCS + LMWH); Test type: Superiority; p < 0.001, Fisher Exact

8. Secondary Outcome: Number of Patients Who Died From VTE at 30 Days After Surgery
Description: VTE related deaths that occurred during inpatients and outpatient period of treatment and were confirmed by autopsy
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group (SCD + GCS + LMWH) | Control Group (GCS + LMWH)
Number analyzed (Participants) | 193 | 194
Participants | 0 | 2

9. Secondary Outcome: Number of Patients With Symptomatic and Asymptomatic VTE Events at 180 Days After Surgery
Description: Taking into account all symptomatic and asymptomatic VTE events confirmed by duplex ultrasound, CTPA, SPECT/CT, autopsy or other appropriate methods of diagnosis that occurred during the inpatient period of treatment and outpatient period of observation
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group (SCD + GCS + LMWH) | Control Group (GCS + LMWH)
Number analyzed (Participants) | 167 | 158
Participants | 1 | 35
Statistical Analysis 1: Comparison: Experimental Group (SCD + GCS + LMWH) vs Control Group (GCS + LMWH); Test type: Superiority; p < 0.001, Fisher Exact

10. Secondary Outcome: Number of Patients Who Died From VTE at 180 Days After Surgery
Description: VTE related deaths that occurred during inpatients and outpatient period of treatment and were confirmed by autopsy
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group (SCD + GCS + LMWH) | Control Group (GCS + LMWH)
Number analyzed (Participants) | 167 | 158
Participants | 0 | 3

11. Other Pre Specified Outcome: Duration of Inpatient Period of Treatment
Description: The inpatient period of treatment suggests time from surgical intervention to discharge from the hospital or death.
Time Frame: time of discharge from the hospital or death, up to 45 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Experimental Group (SCD + GCS + LMWH) | Control Group (GCS + LMWH)
Number analyzed (Participants) | 204 | 203
days | 10 [8 to 12] | 10 [8 to 13]

ADVERSE EVENTS:
Time Frame: 30 days after surgery for most of the adverse events except all-cause mortality that reported over 6 months
Arm/Group | Experimental Group (SCD + GCS + LMWH) | Control Group (GCS + LMWH)
All-Cause Mortality (participants affected / at risk) | 11/204 | 18/203
Serious Adverse Events (participants affected / at risk) | 5/204 | 4/203
Other Adverse Events (participants affected / at risk) | 27/204 | 22/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group (SCD + GCS + LMWH) (N=204) | Control Group (GCS + LMWH) (N=203)
Major bleeding (Blood and lymphatic system disorders) | 5 (5) | 4 (4) — Major bleeding defined by the International Society of Thrombosis and Hemostasis (ISTH) (no enough space to provide full definition from Journal of Thrombosis and Haemostasis, 8: 202-204)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group (SCD + GCS + LMWH) (N=204) | Control Group (GCS + LMWH) (N=203)
Skin hyperemia on lower limbs (Injury, poisoning and procedural complications) | 18 (18) | 13 (13) — Irritation of the skin on lower limbs in the zone of application of GCS and SCD
Skin blisters on lower limbs (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) — Deeper skin injury with the formation of blisters in the zone of application of GCS and SCD
Skin necrosis on lower limbs (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) — Deep lesion of the skin and soft tissues in the zone of application of GCS and SCD
Clinical relevant non-major bleeding (Blood and lymphatic system disorders) | 2 (2) | 7 (7) — Bleeding, that does not match the criteria of major but needs some specific measures for hemostasis and/or interruption or preliminary abortion of anticoagulation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT03044574/Prot_SAP_001.pdf